CLINICAL TRIAL: NCT02394210
Title: Post-authorisation Observational Registry to Assess the Clinical Impact of Initiating Anti-tumour Rescue Therapy in Patients With Multiple Myeloma (MM) in Asymptomatic Biological Relapse Compared to Initiating Treatment at the Time of Symptomatic Relapse.
Brief Title: Post-authorisation Study of Biological Relapse in Patients With Multiple Myeloma
Acronym: EPA-MMBR
Status: Terminated | Type: Observational
Why Stopped: Bias in the study
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-MIE-2012-02
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma asymptomatic relapse symptomatic relapse; IMW Consensus Panel; anti-MM therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients in relapse/biological progression (under the criteria of the IMW (International Myeloma Workshop) Consensus Panel 1 not receiving treatment until clinical relapse.
- Group 2: Patients in relapse/biological progression receiving anti-MM treatment at the time of relapse/biological progression): Patients in this group may receive conventional anti-myeloma treatment as per routine clinical practice at the participating site:
  1. Upon relapse/biological progression, defined as per the criteria of the IMW (International Myeloma Workshop) Consensus Panel Panel1 Or
  2. Upon a significant relapse of paraprotein, defined as:
     * Duplication of M-component in two consecutive readings taken ≤2 months apart; or
     * An increase in absolute levels of serum M-protein ≥1 g/dL or M-protein in urine at ≥500 mg/24h, or
     * Increase in light chain levels ≥20 mg/dL with an abnormal ratio in two consecutive readings taken ≤2 months apart), which suggests the presence of biological progression/relapse criteria, but without including any clinical details of those involved in clinical relapse.

SUMMARY:
Post-authorisation prospective follow-up study to assess the clinical impact on time to progression (TTP) from the start of anti- multiple myeloma treatment at the onset of asymptomatic relapse/biological progression versus start of treatment at the time of symptomatic relapse.

DETAILED DESCRIPTION:
National, observational, prospective, post-authorisation multicentre registry.

It will include patients with a diagnosis of MM who have received no more than two lines of treatment and with at least one partial relapse (≥ PR) with their latest anti-MM treatment, duly documented in accordance with the criteria of the IMW Consensus Panel 1:

1. Patients prior to relapse/biological progression, even without being in asymptomatic relapse/biological progression are followed every one or two months at most, according to the clinical judgment of the physician investigator, and provided there is an analysis (proteinogram and/or immunofixation) in the two months (+/- 15 days) prior to inclusion in which it can be documented that the patient was not in a situation of asymptomatic relapse or progression.

Patients in first or second relapse/biological progression who initiate any of the treatments currently approved and marketed in Spain for the treatment of relapsed MM, based on the criteria of the International Myeloma Workshop (IMW) Consensus Panel 11 or patients without treatment from relapse/biological progression to clinical relapse who initiate treatment after clinical relapse, according to standard criteria for clinical practice, and according to the clinical decision of each participating physician in the study, and provided there is an analysis (proteinogram and/or immunofixation) in the two months (+/- 15 days) prior to inclusion in which it can be documented that the patient was not in a situation of relapse or asymptomatic progression.

Therefore, two groups are defined for inclusion in the registry for patients in 1st or 2nd relapse/biological progression, depending on the treatment strategy adopted according to the routine clinical practice of each site participating in the study.

Group 1: Patients in relapse/biological progression not receiving treatment until clinical relapse.

Relapse/biological progression, under the criteria of the IMW (International Myeloma Workshop) Consensus Panel 11, is understood to be an asymptomatic relapse (without CRAB symptoms) defined by a ≥25% increase over the lowest value obtained during response, in any of the following:

* Serum M-protein (absolute increase must be ≥0.5 g/dL) and/or
* Urine M-component (absolute increase must be ≥200 mg/24 hrs.) and/or
* Only for patients without measurable disease in serum and urine, a 25% increase from the lowest difference in correlated and uncorrelated FLC (absolute increase >10 mg/dL)
* In patients with unmeasurable M-protein in serum and urine, and unmeasurable FLC levels, a 25% increase in the percentage of plasma cells in bone marrow (the absolute percentage must be ≥10%)
* In patients with asymptomatic relapse/biological progression from complete response, recurrence of M protein in serum or urine by immunofixation or electrophoresis in two consecutive samples[1]
* Patients in this group will be studied in two phases:

  * Phase 1 (observation phase): Patients not initially receiving anti-myeloma (anti-MM) treatment, thus patients not treated for myeloma between relapse/biological progression and clinical relapse.
  * Phase 2 (anti-MM treatment after clinical relapse): Patients receive conventional anti-myeloma treatment after clinical relapse*.

Group 2: (anti-MM treatment at the time of relapse/biological progression): Patients in this group may receive conventional anti-myeloma treatment as per routine clinical practice at the participating site:

1. Upon relapse/biological progression, defined as per the criteria of the IMW (International Myeloma Workshop) Consensus Panel Panel1, as an asymptomatic relapse (without CRAB symptoms), defined by a ≥25% increase over the lowest value obtained during remission, in any of the following:

   * Serum M-protein (absolute increase must be ≥0.5 g/dL) and/or
   * Urine M-component (absolute increase must be ≥200 mg/24 hrs.), and/or
   * Only for patients without measurable disease in serum and urine, a 25% increase over the lowest difference in correlated and uncorrelated FLC (absolute increase >10 mg/dL)
   * In patients with unmeasurable M-protein in serum and urine, and unmeasurable FLC levels, a 25% increase in the percentage of plasma cells in bone marrow (the absolute percentage must be ≥10%)
   * In patients with asymptomatic relapse/biological progression from complete response, recurrence of M protein in serum or urine by immunofixation or electrophoresis in two consecutive samples[1] Or
2. Upon a significant relapse of paraprotein, defined as:

   * Duplication of M-component in two consecutive readings taken ≤2 months apart; or
   * An increase in absolute levels of serum M-protein ≥1 g/dL or M-protein in urine at ≥500 mg/24h, or
   * Increase in light chain levels ≥20 mg/dL with an abnormal ratio in two consecutive readings taken ≤2 months apart), which suggests the presence of biological progression/relapse criteria, but without including any clinical details of those involved in clinical relapse*.

     * any change in treatment regimens, for example, discontinuation or addition of a drug (except changes in dose for any of the initial drugs) will mark the end of the anti-MM treatment phase and passing of the patient to the 36-month post-treatment follow-up phase.

In case of temporary interruptions of the study drug, under 30 days, or of any duration (except if the reason for the interruption is toxicity, the patient will continue in the anti-MM treatment phase, provided the same treatment regimen is resumed.

Patients included in the registry prior to relapse/biological progression, will be assigned to group 1 or 2 according to the strategy that the investigator decides once relapse/biological progression occurs. Furthermore, to include these patients in the phase prior to relapse/biological progression there must be an analysis (proteinogram and/or immunofixation) in the two months (+/- 15 days) prior to inclusion in which it can be documented that the patient was not in a situation of relapse or asymptomatic progression.

If patients included in the registry stage prior to relapse/biological progression relapse or progress directly with CRAB criteria they will be considered non-evaluable for the purposes of sample size, although they will be evaluated for the purposes of the secondary exploratory objective defined in section 5.2. In that case, these patients will receive anti-MM treatment/s for recurrence or progression according to clinical practice in the participating sites.

Likewise, patients who after being included in the registry receive treatment within a clinical trial will be deemed not evaluable.

From the time relapse/biological progression occurs, the investigator shall have a period of two months to decide in which observation group to include the patient.

Follow-up is established for the duration of the anti-MM treatment phase. For all patients included in the registry and whenever possible, the prospective follow-up period will be extended an additional 36 months (data collected every 6 months), starting this phase from the last dose of study medication.

Once patients have been included on the registry, they must be followed at a maximum of two month intervals, until relapse or progression of the disease, with the inclusion of data in the electronic case report form every 2 months (for patients included in the registry after relapse/biological progression), or every 4 months (for patients included in the registry prior to relapse/biological progression), in order to allow an exact calculation of TTP (primary endpoint) and the time from relapse/biological progression to clinical relapse.

To this end, the proteinogram and/or immunofixation (in case of negative protein count) must have been assessed every one or two months during or after completion of treatment prior to inclusion.

However, given the observational nature of the study, patient follow-up will take place as per routine clinical practice at each site.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, greater than or equal to 18 years of age patients with a diagnosis of Multiple Myeloma (MM) based on the international criteria.
2. Patients with a diagnosis of Multiple Myeloma who had not received more than two regimen therapies and who had achieved at least a Partial Response (PR) with the last anti- Multiple Myeloma treatment according the criteria of the IMW (International Myeloma Workshop) Consensus Panel 1, included before relapse/biological progression or with an asymptomatic relapse (without Calcium increase, Renal Impairment, Anemia and Bone Lesion (CRAB) symptoms) defined by a ≥25% increase on the lowest value obtained during remission, in any of the following:

   * Serum M-protein (absolute increase must be ≥05 g/dL) and/or
   * Urine M-component (absolute increase must be ≥ 200 Mg/24 hrs.), and/or
   * Only for patients without measurable components in serum and urine, a 25% increase on the lowest difference in Free light chain (FLC) ratios (absolute increase >10 mg/dL)
   * In patients with unmeasurable M-protein in serum and urine, and unmeasurable FLC levels, a 25% increase in the percentage of plasma cells in bone marrow (the absolute percentage must be ≥10%) In any case, it is necessary to have an analysis (proteinogram and/or immunofixation) in the two months (+/- 15 days) prior to inclusion in which it can be documented that the patient was not in a situation of relapse or asymptomatic progression.

   Patients with an asymptomatic relapse/progression from a Complete Response (CR):
   * Reappearance of serum or urine M-protein by immunofixation or electrophoresis
3. Patients who consent in writing after they has clearly explained the nature and purpose of the study (consent written informed).

Exclusion Criteria:

1. Patients who are participating in an interventional clinical trial.
2. Patients that refuse to participate in the study.
3. Patients who present physical or mental incapacity to understand the information that is supplied, and/or respond to questions their doctor will perform as part of the study.
4. Clinical Relapse Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of MM having received first or second-line treatment who have achieved ≥PR since their last anti-MM treatment, so that patients may be included in the registry before relapse/biological progression while followed every 1 to 2 months based on routine clinical practice, as well as at the time relapse/biological progression is detected, as per the criteria of the IMW Consensus Panel 11.
Sampling Method: Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | Up to 38 months
  The period from when relapse/biological progression is detected until a new relapse or progression of tumour to the treatment received for biological or clinical relapse is documented according to the criteria of the IMW Consensus Panel.

SECONDARY OUTCOMES:
Race of participants at Baseline | Baseline visit
  To describe the demographic characteristics of patients with multiple myeloma (MM) in relapse/biological progression.
Age of participants at Baseline | Baseline visit
  To describe the demographic characteristics of patients with MM in relapse/biological progression.
Gender of participants at Baseline | Baseline visit
  To describe the demographic characteristics of patients with MM in relapse/biological progression.
Stage of Multiple Myeloma (MM) before study entry based on the international staging system (ISS) | Baseline visit
  Providing the stages of MM based on the international staging system (ISS)
Time from first pathologic diagnosis | Baseline visit
  Time from initial diagnosis to the first pathological fracture in patients with MM
The number of Comorbidities | Baseline visit
  The incidence of comorbidities associated with patients with MM
Concomitant treatments related to MM | Baseline visit
  The type of medication/treatment that the patients have received for MM patients
ECOG performance status | Baseline visit
  To define the Eastern Cooperative Oncology Group (ECOG) performance status at the base line visit only
Define the abnormal finding in complete blood count at base line | Baseline visit
  To define the number of abnormal findings in hematology panel at baseline.
Define the abnormal findings within the Biochemistry panel | Baseline visit
  To define number of abnormal findings within the Biochemistry panel at baseline.
The time from biological progression until clinical relapse | Up to 38 months
  To assess the median time elapsing from biological progression until clinical relapse in patients with MM who do not receive treatment until clinical relapse as per the criteria of the IMW Consensus Panel 11
Overall Response rate | Up to 38 months
  To assess the overall response rate for the different anti-myeloma treatments as per the uniform criteria of the IMW Consensus Panel 11.
Event-free survival (EFS) | Up to 38 months
  Is from baseline to the appearance of the event; considering as an event symptomatic relapse, progression or death.
Progression-free survival (PFS) | Up to 38 months
  Is from baseline to the appearance of the event; considering as an event tumor progression or death from any cause.
Overall survival (OS) | Up to 38 months
  Is measured from symptomatic relapse until death from any cause
EORTC QLQ-C30 Questionnaire | Up to 38 months
  Is European Organization for Research and Treatment of Cancer, specifically for the assessment of quality of life in cancer patients.
QLQ-MY24 Questionnaire | Up to 38 months
  Questionnaire QLQ-MY24 addresses four areas of quality of life important in MM: a pain scale, side effects of treatment, social support and future perspective.
Cost associated with participants visit to hospital/primary health care associated with anti-myeloma therapy | Up to 38 months
  To describe the costs associated with therapy for MM in clinical practice that are measurable from a financial perspective and to explore the differences between the different treatment regimens administered under the study. This includes, visits to hospital/primary health care center.
Adverse Events (AEs) | Up to 38 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mireya Navarro, MD, Study Director — Celgene
Locations (44):
- Spain (44):
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Royo Villanova, Zaragoza, Aragon
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital de Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Txagorritxu, Vitoria-Gasteiz, Basque Country
  - Hospital Universitario de Canarias, La Laguna. Santa Cruz de Tenerife, Canary Islands
  - Hospital de Gran Canaria, Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Ntra. Sra. de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Marqués de Valdecilla, Santander, Cantabria
  - Hospital Nuestra Señora de Sonsoles Avila, Ávila, Castille and León
  - Hospital de Burgos, Burgos, Castille and León
  - Hospital de León, León, Castille and León
  - Hospital de Segovia, Segovia, Castille and León
  - Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Vall d´Hebron, Barcelona, Catalonia
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Josep Trueta de Girona, Girona, Catalonia
  - Hospital Arnau de Vilanova de Lleida, Lleida, Catalonia
  - Hospital de Sabadell ( Parc Taulí), Sabadell, Catalonia
  - Complejo Hospitalario de Cáceres (S. Pedro de Alcántara), Cáceres, Extremadura
  - Hospital de Llerena, Llerena, Badajoz, Extremadura
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Complexo Hospitalario de Ourense, Ourense, Galicia
  - Hospital Montecelo, Pontevedra, Galicia
  - Complejo Hospitalario Universitario de Vigo, Vigo, Galicia
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Quirón, Pozuelo de Alarcón, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Santa Lucía, Cartagena, Murcia
  - Hospital Virgen de Arrixaca, El Palmar, Murcia, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General de Castellon, Catellón, Valencia
  - Hospital Clínico Universitario Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova (Valencia), Valencia, Valencia
  - Hospital de Manises, Valencia, Valencia
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Infanta Leonor, Madrid
  - Complejo Universitario de San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid